CLINICAL TRIAL: NCT05305014
Title: Contribution of Inflammation and Neuronal Integrity Markers in Patients With First-episode Conversive Motor Disorder
Acronym: HYCOIN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2021/IC-01
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2023-05

CONDITIONS: Conversion Disorder
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with conversive motor disorder: Patients with paralysis, motor weakness or abnormal movements meeting the DSM-IV criteria of conversive motor disorder consulting the SAU or the Neurology departments of the CHU of Nîmes and Montpellier included in the HYCORE parent study (RCB ID 2014-A01159-38, NCT02329626)
  Interventions: Diagnostic Test: blood inflammatory markers (TNF-α, IL1ra, RsIL-2, IL-6, IL-10, IL-18, IFNγ, MCP-1/CCL2 GFAP)

INTERVENTIONS:
Diagnostic Test: blood inflammatory markers (TNF-α, IL1ra, RsIL-2, IL-6, IL-10, IL-18, IFNγ, MCP-1/CCL2 GFAP) — Bioassays of blood inflammatory markers (TNF-α, IL1ra, RsIL-2, IL-6, IL-10, IL-18, IFNγ, MCP-1/CCL2 GFAP) from sera babcocked in the HYCORE mother study.

SUMMARY:
Conversion disorders, also called "dissociative disorders" (ICD-10), or "functional neurological disorders" (DSM-5), are a common condition, with a prevalence of 1-10% in medical and surgical inpatients (Toone 1990), and 10-30% in neurology patients (Carson et al. 2000).

They are characterized by the presence of symptoms or deficits affecting voluntary motor, sensory, or sensory functions suggestive of a neurological or general medical condition in combination with psychological factors. Functional neurological disorder is currently a diagnosis of elimination and its treatment remains uncodified. A better understanding of the pathophysiology of this disorder is needed to improve the diagnostic and therapeutic approach to this condition.

Identifying new biological markers associated with motor symptoms occurring during the course of the functional neurological disorder would allow clinicians to acquire new diagnostic methods, to improve therapeutic means and their specificity and to highlight possible predictive factors of the clinical evolution of this pathology. At the same time, the identification of biological markers associated with motor symptoms will allow the patient to better understand and accept the diagnosis, and thus to better adhere to the proposed treatment.

DETAILED DESCRIPTION:
This project is an ancillary study carried out from the cohort of patients included in the HYCORE protocol "PET-Scan evaluation of metabolic abnormalities associated with the clinical evolution at 6 months of patients suffering from a motor conversion disorder" (RCB N°: 2014-A01159-38) of which the CHU of Nîmes is the promoter. In the HYCORE project, 20 patients suffering from a first episode of motor conversion disorder (with paralysis, motor weakness or abnormal movements according to DSM-IV criteria) in acute phase (evolving for less than one month) recruited in the neurology and psychiatry departments of the University Hospital of Montpellier and Nîmes are included.

Thinvestigtor plan to use the biological samples collected in the HYCORE project for the determination of markers of inflammation and neurofilaments (GFAP & NfL); the levels of inflammatory markers thus obtained will be put into perspective in relation to the cerebral metabolism observed by PET-scan as well as the persistence of a motor handicap (EDSS score) evaluated in the HYCORE study.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given free and informed consent and signed the consent.
* Patient must be enrolled in or a beneficiary of a health insurance plan.
* Patient's age is > 18 and ≤ 65 years.
* Patient meets DSM-IV criteria for conversive motor disorder (with paralysis, motor weakness, or abnormal movements) evolving for less than 1 month and is euthymic (HAMD score < or =7 assessed by a psychiatrist).
* First episode (incident case)
* The last symptom is less than one month old.
* The patient is not on neuroleptics.

Exclusion Criteria:

* Subject is participating in another study
* Subject is in an exclusion period determined by a previous study
* Subject is under court protection, guardianship, or conservatorship
* The subject refuses to sign the consent form
* It is impossible to provide the subject with informed information
* The patient is pregnant, parturient, or nursing
* Specialized neurological clinical examination and brain and spinal cord MRI reveal organic neurological damage
* The subject presents a HAMD score >7
* Subject has a current manic or hypomanic episode, a current diagnosis of substance abuse/dependence (excluding tobacco), a lifetime diagnosis of schizophrenia, or a chronic neurological condition (active epilepsy, stroke, brain tumor)
* Suicidal or high-risk subjects (assessed using the MINI)
* The subject has a contraindication to the performance of a PET scan
* Patient is on neuroleptic medication at inclusion
* The last symptom is more than one month old
* The patient has already had an episode (prevalent case).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients with paralysis, motor weakness or abnormal movements corresponding to the DSM-IV criteria of conversive motor disorder consulting the SAU or the Neurology departments of the CHU of Nîmes and Montpellier already included in the HYCORE mother study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
TNF-α | Baseline
  Correlation between blood TNF-α and resting metabolic abnormalities on 18-FDG PET scan in the acute phase of a first episode of conversive motor disorder.
IL1ra | Baseline
  Correlation between blood IL1ra and resting metabolic abnormalities on 18-FDG PET scan in the acute phase of a first episode of conversive motor disorder.
RsIL-2 | Baseline
  Correlation between blood RsIL-2 and resting metabolic abnormalities on 18-FDG PET scan in the acute phase of a first episode of conversive motor disorder.
IL-6 | Baseline
  Correlation between blood IL-6 and resting metabolic abnormalities on 18-FDG PET scan in the acute phase of a first episode of conversive motor disorder.
IL-10 | Baseline
  Correlation between blood IL-10 and resting metabolic abnormalities on 18-FDG PET scan in the acute phase of a first episode of conversive motor disorder.
IL-18 | Baseline
  Correlation between blood IL-18 and resting metabolic abnormalities on 18-FDG PET scan in the acute phase of a first episode of conversive motor disorder.
IFNγ | Baseline
  Correlation between blood IFNγ and resting metabolic abnormalities on 18-FDG PET scan in the acute phase of a first episode of conversive motor disorder.
MCP-1/CCL2 | Baseline
  Correlation between blood MCP-1/CCL2 and resting metabolic abnormalities on 18-FDG PET scan in the acute phase of a first episode of conversive motor disorder.
GFAP | Baseline
  Correlation between blood GFAP and resting metabolic abnormalities on 18-FDG PET scan in the acute phase of a first episode of conversive motor disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- Ismael CONEJERO, Nîmes, Choisir Une Région, France

REFERENCES:
- [Result] Conejero I, Thouvenot E, Hingray C, Hubsch C, El-Hage W, Carle-Toulemonde G, Rotge JY, Drapier S, Drapier D, Mouchabac S. [Understanding functional neurological disorders: From biological markers to pathophysiological models]. Encephale. 2023 Aug;49(4S):S18-S23. doi: 10.1016/j.encep.2023.06.003. Epub 2023 Jul 1. French. PMID 37394415